CLINICAL TRIAL: NCT06772909
Title: Prevalence Of Renal Dysfunction In Patients With Chronic Liver Disease Admitted To Sohag University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Hossam Mohamed, Resident doctor, Sohag University
Other Study IDs: Soh-Med--24-12-10MS
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Renal Dysfunction
MeSH Terms: conditions — Renal Insufficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — no intervention

SUMMARY:
To find out the prevalence of renal dysfunction in chronic liver disease patients who admitted to sohag university hospital

DETAILED DESCRIPTION:
The interrelationship between liver disease and renal dysfunction was recognized as early as the era of Hippocrates and this has been the object of a considerable amount of research since then. Kidney dysfunction in liver disease can be due to different etiologies and can have diverse manifestations. Most of the abnormalities of kidney function in cirrhosis are of functional origin- namely, sodium retention, impaired free water excretion, and renal vasoconstriction with a decrease in renal perfusion and glomerular filtration rate.

Renal dysfunction in chronic liver disease usually follows a progressive course - the final phase being Hepatorenal syndrome (HRS).

There is no explanation that fully defines the complex relationship between the diseased liver and disturbances in kidney function, though substantial progress is being made in recent years regarding research in this aspect. One of the most difficult issues in the clinical evaluation of patients with cirrhosis is the accurate assessment of renal function. Standard measures of renal function like blood urea nitrogen and serum creatinine are likely to give erroneous impressions and hence alternative methods to determine renal reserve must be used.

Kidney function is evaluated by assessing the glomerular filtration rate (GFR) For many years now, the assessment of GFR has relied on the measurement of the concentration of serum creatinine, which is associated with many problems. Creatinine is a product of the metabolism of creatine, produced in the liver from three amino acids, methionine, arginine, and glycine, and stored in muscle to be used as a source of energy once phosphorylated. Creatinine does not appear in the plasma at a constant rate; it is secreted in the tubule and can undergo extrarenal elimination, thought to involve creatinase in the gut. Serum creatinine concentration displays an exponential relationship with GFR, rendering it specific, but not a sensitive measure of GFR. The creatinine pool is affected by gender, age, ethnicity, nutritional state, protein intake, and importantly liver disease. 1 In chronic liver disease, the reduction in the serum creatinine pool is due to a 50% decrease in hepatic production of creatine; increases in the volume of distribution due to the accumulation of extracellular fluid, edema, and ascites; malnutrition and loss of muscle mass, which is related to repeated episodes of sepsis and large-volume ascites affecting satiety.2 Ultimately, patients with chronic liver disease have a significantly lower baseline serum creatinine concentration than the general population (35-75 μmol/l).

Patients with chronic liver disease display smaller and delayed (up to 48-72 hours) changes in serum creatinine for a given change in GFR, thus impairing the recognition and underestimating the degree of change in GFR.3,4 Detection of renal insufficiency is clinically important because it contributes significantly to high morbidity and mortality in cirrhosis. Moreover, renal dysfunction is one of the most important risk factors when liver transplantation is being considered. Patients with cirrhosis and renal failure are at high risk for death while awaiting transplantation and have an increased frequency of complications and reduced survival after transplantation, as compared with those without renal failure.

ELIGIBILITY:
Inclusion Criteria:

- Data regarding demographic variables (age, weight, sex),

Evidence for chronic liver disease is defined by:

A compatible Clinical profile (signs of liver cell failure or reduced liver span) along with Biochemical (altered liver function tests, reversal of albumin globulin ratio, etc) or Sonographic evidence (altered echotexture of the liver) Diuretics will be withheld for 3 days before carrying out lab investigations.

Exclusion Criteria:

* • patients >70 years

  * Known primary renal disease or obstructive uropathy
  * Diabetes mellitus
  * Hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prevalence of renal dysfunction in chronic liver disease patients who admitted to sohag university hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of renal dysfunction in patients with chronic liver disease | during admission time at sohag university hospital
  prevalence of renal dysfunction in patients with chronic liver disease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.proquest.com/pqdtglobal1/dissertations-theses/renal-function-chronic-liver-disease/docview/2866353338/sem-2?accountid=178282